CLINICAL TRIAL: NCT07381764
Title: ROMANCE GOIM Study: A Phase II, Open Label, Multicenter Trial Investigating Irinotecan Plus Cetuximab Rechallenge Compared With Trifluridine/Tipiracil Plus Bevacizumab as Third Line Treatment in Circulating Tumor DNA Molecularly Selected Metastatic Colorectal Cancer
Brief Title: ROMANCE: "Irinotecan Plus Cetuximab Rechallenge Versus Trifluridine/Tipiracil Plus Bevacizumab in Molecularly Selected Metastatic Colorectal Cancer"
Acronym: ROMANCE - GOIM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italia Meridionale (Other)
Responsible Party: Principal Investigator, Davide Ciardiello, Principal Investigator, Gruppo Oncologico Italia Meridionale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROMANCE - GOIM; 2025-521319-38-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab; Irinotecan; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: ARM A: Cetuximab + irinotecan (75 patients) ARM B: Trifluridine/tipiracil + bevacizumab (75 patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Arm A - Irinotecan + Cetuximab (Experimental): This arm is for participants with molecularly selected metastatic colorectal cancer who have progressed after standard first- and second-line therapies and previously achieved clinical benefit from an anti-EGFR-based regimen. Participants randomized to this arm will receive irinotecan in combination with cetuximab as a rechallenge strategy. The objective of this arm is to evaluate the antitumor activity and safety of irinotecan plus cetuximab compared with the control treatment in the third-line setting.
  Interventions: Drug: Erbitux (Cetuximab); Drug: Irinotecan
- Active Comparator: Arm B - Trifluridine/Tipiracil + Bevacizumab (Active Comparator): This arm is for participants with molecularly selected metastatic colorectal cancer who have progressed after standard first- and second-line therapies. Participants randomized to this arm will receive trifluridine/tipiracil in combination with bevacizumab, which represents the current standard of care in the third-line treatment setting. This arm serves as the control group for comparison with the experimental rechallenge strategy.
  Interventions: Drug: Bevacizumab; Drug: Trifluridine/tipiracil

INTERVENTIONS:
Drug: Erbitux (Cetuximab) — This is an anti-EGFR monoclonal antibody administered in combination with chemotherapy. The dose is 500 mg/m2 over 120 minutes
  Arms: Experimental: Arm A - Irinotecan + Cetuximab
Drug: Bevacizumab — This is an anti-VEGF monoclonal antibody used as an active comparator in the control arm of the study. The dose is 5 mg/Kg of body weight given once every 2 weeks.
  Arms: Active Comparator: Arm B - Trifluridine/Tipiracil + Bevacizumab
Drug: Irinotecan — Irinotecan is a cytotoxic chemotherapy agent administered intravenously in combination with cetuximab the dose is 180 mg/m2 over 90 minutes, once every 2 weeks.
  Arms: Experimental: Arm A - Irinotecan + Cetuximab
Drug: Trifluridine/tipiracil — Trifluridine/tipiracil is an oral antineoplastic combination administered in combination with bevacizumab as part of the control treatment arm. The dose is 5 mg/ m² twice daily on Days 1 to 5 and Days 8 to 12 on a cycle of 28 days.
  Arms: Active Comparator: Arm B - Trifluridine/Tipiracil + Bevacizumab

SUMMARY:
This study is a phase II, open-label, multicenter clinical trial designed to evaluate two different treatment options for patients with metastatic colorectal cancer whose disease has progressed after standard therapies. The study compares a rechallenge treatment using irinotecan plus cetuximab with the current standard of care, trifluridine/tipiracil plus bevacizumab, as third-line therapy. Patients enrolled in the study are selected based on specific molecular characteristics of their cancer, identified through circulating tumor DNA analysis from a blood sample. The main purpose of the study is to determine whether the rechallenge with irinotecan and cetuximab leads to a higher tumor response rate compared with trifluridine/tipiracil plus bevacizumab. Secondary objectives include evaluating progression-free survival, overall survival, safety, and quality of life. Patients will be randomly assigned to one of the two treatment groups and will receive treatment until disease progression, unacceptable side effects, or withdrawal of consent. Tumor response will be assessed using standard imaging techniques according to RECIST criteria.

DETAILED DESCRIPTION:
This is a phase II, open-label, randomized, multicenter clinical trial designed to evaluate the efficacy and safety of an anti-EGFR rechallenge strategy compared with the current standard of care in patients with molecularly selected metastatic colorectal cancer (mCRC). Eligible patients have metastatic colorectal cancer that has progressed after standard first- and second-line therapies and have previously achieved clinical benefit from an anti-EGFR-based regimen. Patient selection is based on molecular profiling performed on circulating tumor DNA obtained from a baseline blood sample, identifying tumors that are wild-type for RAS, BRAF, EGFR, PIK3CA exon 20, MAP2K1, and MET, and without HER2 amplification. A total of 150 patients will be randomized in a 1:1 ratio to one of two treatment arms. In the experimental arm, patients will receive cetuximab in combination with irinotecan administered every two weeks. In the control arm, patients will receive trifluridine/tipiracil administered orally according to standard dosing schedules in combination with bevacizumab administered every two weeks. Treatment in both arms will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other protocol-defined discontinuation criteria. Tumor assessments will be performed at regular intervals using computed tomography or magnetic resonance imaging and evaluated according to RECIST version 1.1 criteria. The primary endpoint of the study is the objective response rate. Secondary endpoints include progression-free survival, overall survival, safety and tolerability, and quality of life assessed using validated questionnaires. Adverse events will be monitored throughout the study and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0. Following disease progression, crossover to the alternative treatment arm may be considered at the investigator's discretion. Long-term follow-up will be conducted to assess survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years
2. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) ≤1
3. Diagnosis of histologically or cytologically confirmed colorectal cancer.
4. At least one measurable lesion according to RECIST1.1
5. KRAS/NRAS/BRAFV600E wt status of primary CRC or related metastasis (local laboratory assessment).
6. Progression to previous first-line anti-EGFR-containing therapy producing at least a partial response ≥ 6 months.
7. Received and progressed to an anti-EGFR and irinotecan free second-line treatment.
8. Have an anti-EGFR free interval of at least 4 months.
9. Refractory to previous 5-fluorouracil/capecitabine, irinotecan, oxaliplatin, bevacizumab.
10. RAS/BRAF/EGFR/PIK3CAex20/MAP2K1/MET WT and HER2 not amplified ctDNA at FoundationOne CDx test at baseline.
11. Life expectancy of at least 3 months.
12. Adequate hematological function defined by white blood cell (WBC) count ≥ 2.5 × 109/L with absolute neutrophil count (ANC) ≥ 1.5 × 109/L, lymphocyte count ≥ 0.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused).
13. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and alanine aminotransferase (ALT) levels ≤ 2.5 × ULN for all subjects or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
14. Adequate renal function defined by an estimated creatinine clearance > 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
15. No contraindication to the study drugs.
16. No prior treatment with trifluridine/tipiracil.
17. Women of childbearing potential* must have a negative blood pregnancy test at thescreening visit. Subjects and their partners must be willing to avoid pregnancy during the trial.

    *A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
18. Women of childbearing potential, or male, must agree to use adequate contraception (e.g., abstinence, intrauterine device, oral contraceptive, or double-barrier method), during the study and until at least 6 months after last dose of study treatment administration, based on the judgment of the Investigator or a designated associate.
19. Will and ability to comply with the protocol.
20. Signed informed consent obtained before screening.

Exclusion Criteria:

1. ECOG PS ≥2
2. Received more than 2 lines of treatment for metastatic disease.
3. Previous treatment with trifluridine/tipiracil
4. RAS/BRAF/EGFR/PIK3CAex20/MAP2K1/MET WT HER2 not amplified status at liquid biopsy analysis during screening.
5. Previous history of malignancy within the last 2 years will be excluded with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ
6. Evidence of bleeding diathesis or coagulopathy.
7. Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.
8. Known severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 5 Grade ≥ 3), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).
9. Clinically significant cardiovascular disease, active inflammatory bowel disease, active autoimmune disease.
10. Diagnosis of interstitial pneumonitis or pulmonary fibrosis.
11. History of abdominal fistula, GI perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to the first study treatment.
12. Pregnant or lactating women.
13. Psychiatric or addictive disorders would preclude study participation.
14. Active uncontrolled infections or other clinically relevant concomitant illness contraindicating study treatments.
15. Withdrawal of the consent to take part to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2031-03-30 (Estimated); Study Completion 2031-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From Week 8 through disease progression or end of treatment, up to approximately 24 months.
  Objective Response Rate (ORR) is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria. Tumor assessments are based on radiological imaging reviewed centrally by an independent blinded radiology reviewe

SECONDARY OUTCOMES:
Progressio-Free Survival (PFS) | From date of randomization until the date of first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first, assessed up to 36 months.
  Progression-Free Survival (PFS) is defined as the time from randomization to documented disease progression according to RECIST version 1.1 criteria or death from any cause, whichever occurs first.
Overall Survival (OS) | From date of enrollment until death from any cause, assessed up to 36 months.
  Overall Survival (OS) is defined as the time from enrollment to death from any cause.
Incidence of Adverse Events and Serious Adverse Events | From first dose of study treatment until 30 days after the last dose of study treatment.
  Safety will be assessed by the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), as well as by changes in clinical laboratory parameters, vital signs, physical examinations, electrocardiogram (ECG) findings, and ECOG performance status. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Treatment Exposure as a Measure of Tolerability | Through study completion, an average of approximately 24 months
  Tolerability will be assessed by the frequency of treatment discontinuations, dose reductions, and dose delays due to adverse events during study treatment.
The impact of treatment with irinotecan plus cetuximab and trifluridine/tipiracil plus bevacizumab on quality of life | From baseline through study completion, an average of approximately 12 months
  The impact of treatment with irinotecan plus cetuximab and trifluridine/tipiracil plus bevacizumab on quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).

OTHER OUTCOMES:
Progression-Free Survival (PFS) of the Subsequent Line of Treatment | From initiation of subsequent line of treatment until documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first, assessed up to approximately 36 months.
  Progression-Free Survival (PFS) following the subsequent line of treatment is defined as the time from initiation of the first subsequent anticancer therapy to the first documented disease progression according to RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (26):
- Italy (26):
  - Azienda Ospedaliero Universitaria "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - A.O.U. Ospedali Riuniti, Ancona
  - Centro di Riferimento Oncologico (CRO), IRCCS, Aviano
  - A.O.R.N. "Sant'anna e San Sebastiano", Caserta
  - Ospedale IRCCS 'Saverio de Bellis', Castellana Grotte
  - A.R.N.A.S. Garibaldi - P.O. Garibaldi-Nesima, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - A.O.U. Careggi, Florence
  - Istituto Romagnolo per lo Studio dei Tumori 'Dino Amadori', Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Casa di Cura Villa Maria, Mirabella Eclano
  - AOU Policlinico di Modena, Modena
  - A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - Istituto Nazionale Tumori 'Fondazione G. Pascale', Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - ARNAS Civico - Di Cristina-Benfratelli - P. O. 'Civico e Benfratelli', Palermo
  - Casa di cura Macchiarella, Palermo
  - A.O.U. Pisana, Pisa
  - Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS, Roma
  - Fondazione IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - A.O.U. Sassari, Sassari
  - Ospedale San Giuseppe Moscati, Statte
  - A.O. 'Pia Fondazione Cardinale G. Panico', Tricase
  - ASST Sette Laghi-Ospedale di Circolo Fondazione Macchi, Varese

IPD SHARING:
Plan to Share IPD: Undecided